CLINICAL TRIAL: NCT05834231
Title: Efficacy of Memantine in Prevention of Oxaliplatin-induced Peripheral Neurotoxicity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Drug: Memantine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — oral
  Arms: Intervention
Drug: Placebo — oral
  Arms: Control

SUMMARY:
Memantine is a drug for the management of Alzheimer's Disease (AD) due to its promising neuroprotective properties. We hypothesize that Memantine possesses a beneficial role against chemotherapy-induced neuronal damages.

ELIGIBILITY:
Inclusion Criteria:

histologically confirmed diagnosis of stage III colorectal cancer performance status < 2 according to Eastern Cooperative Oncology Group (ECOG) score adequate renal function (glomerular filtration rate ≥ 90)

Exclusion Criteria:

preexisting neuropathic or brain disorders, a previous use of chemotherapeutic agents including oxaliplatin use of drugs reported to have neuroprotective role

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced-peripheral neuropathy using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | 6 months

IPD SHARING:
Plan to Share IPD: Undecided